CLINICAL TRIAL: NCT03854630
Title: Hepatitis B Virus Vaccination in HIV-positive Patients and Individuals at High Risk for HIV Infection: an Open-label Randomized Clinical Trial
Brief Title: Hepatitis B Virus Vaccination in HIV-positive Patients and Individuals at High Risk for HIV Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201608051MIPC
Record Dates: First submitted 2017-09-07; First posted 2019-02-26 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Viral Hepatitis B; Immunization; Infection; HIV Infections
MeSH Terms: conditions — Hepatitis B; Infections; HIV Infections | interventions — Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dose (20µg) (Active Comparator): Three doses of 20µg HBV vaccine given intramuscularly at week 0, 4, 24.
  Interventions: Drug: Engerix-B
- Double dose (40µg) (Experimental): Three doses of 40µg HBV vaccine given intramuscularly at week 0, 4, 24.
  Interventions: Drug: Engerix-B

INTERVENTIONS:
Drug: Engerix-B — The vaccine contains HBsAg which was produced by genetic engineering yeast. It stimulates the active immunity generated by human immune system toward the HBsAg.

SUMMARY:
The primary aim of this open-label, randomized control trial is to compare the immunogenicity at week 28 after 20µg HBV vaccine (at week 0, 4, 24) versus 40µg HBV vaccine (40-µg at week 0, 4, 24 week) among HIV-positive patients or HIV-negative MSM who were born in Taiwan after July 1986 and tested negative for all HBV serological markers. The secondary aims are to assess the safety of double-dose HBV vaccination, the proportions of high-level responders (anti-HBs antibody >100 mIU/ml) at weeks 28 and 48, the serological responses at week 48, and incident HBV infection (indicated by appearance of anti-HBc and/or HBsAg) at week 48.

DETAILED DESCRIPTION:
I. Study procedures:

1. Well explain, complete inform and consent documents
2. A blood test for hepatitis B surface antigen (HBsAg), anti-hepatitis B surface antibody (anti-HBs antibody), anti-hepatitis B core antibody (anti-HBc antibody), anti-HCV and RPR will be performed first.
3. The patients with all negative seromarkers (within 1 month) will be allocated to two groups (random blank=4), a standard-dose booster of 20µg and a double-dose booster of 40µg. For patients receiving 40µg, two 20µg of vaccines are injected at both sides of deltoid muscles. The schedules of booster vaccination are the same in two groups, which is at 0, 1, 6 months.
4. To detect and manage possible immediate and severe allergic reaction, patients who received vaccination will be observed for 30 minutes after injection.
5. The solicited adverse effect will be recorded on the diary card if occurred in 7 days after each dose of vaccination.
6. The titer of hepatitis B surface antibody will be examined before booster vaccination, at the 4th week, the 24th week, 28th week, 48th week. By comparing the responses in the two groups, the effect of different doses of booster vaccination can be evaluated. For those HIV-negative individuals at baseline, HIV screening test will be evaluated every 6 months during the study, at the 24th week, the 48th.
7. To screen the acquisition of hepatitis B, the anti-HBc antibody and HBsAg will be examined at the 48th week
8. To screen the acquisition of hepatitis C and syphilis, anti-HCV and RPR will be examined at the 24th week, the 48th week
9. The results of the study will be informed by phone or the physician during the follow-up care.
10. The serum/blood samples will be preserved in the research lab of the department of internal medicine and kept for 20 years. During this period, the sample will be applied or used in other studies after the patients and the Research Ethics Committee both agreed.
11. During the follow-up care, the treatment or record of hospitalization will be recorded or reviewed.
12. The participants will drop out of clinical trial when protocol violation occurred or the participant is not willing to continue.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men (MSM)
* Birth date after 1986/7/1 and aged 20 years or older
* Seronegative for HBsAg, anti-HBs (<10 mIU/ml), and anti-HBc at screening (within 1 month of the first dose)
* Regularly receiving HIV care for HIV-positive patients over the past 6 months
* Seeking VCT for at least once for HIV-negative patients over the past 12 months

Exclusion Criteria:

* Active infection or malignancy within 12 months of screening
* Receiving chemotherapy, immunosuppressant, or IVIG within 12 months of screening
* Received higher than 5 mg of prednisolone, including IV, oral, or topical form, per day for more than 1 weeks within 6 months of screening
* Receiving HBV vaccination within 1 months of screening, or being allergic to HBV vaccine
* Receiving other vaccination within 1 months of screening, such as influenza, pneumococcus, HPV, HAV, varicella vaccine.
* Stage 4 and 5 of chronic kidney disease (GFR<30 mL/min/1.73m), or receiving dialysis.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 575 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaccine efficacy | week 28
  The proportion of patients with Anti-HBs antibody higher than 10mIU/ml

SECONDARY OUTCOMES:
High-titer response | week 28
  The proportion of patients with Anti-HBs antibody higher than 100mIU/ml
Long-term efficacy | 48 weeks
  The proportion of anti-HBs antibody titers higher than 10mIU/ml
Long-term high-titer response | 48 weeks
  The proportion of anti-HBs antibody titers higher than 100mIU/ml
Hepatitis B incident infection rate | 48 weeks,
  new HBsAg and anti-HBc antibody seroconversion
Hepatitis C infection and syphilis infection rate | at 24 week, 48 weeks
  new hepatitis C infection and syphilis infection
HIV seroconversion among HIV-negative MSM | at 24 weeks, 48 weeks
  new HIV seroconversion among HIV-negative MSM

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, MD, PhD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No